CLINICAL TRIAL: NCT02868658
Title: Incidence of Symptomatic and Asymptomatic Influenza Among Healthcare Workers : A Multicenter Cohort Study
Brief Title: Asymptomatic Flu Project
Acronym: AFP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 69HCL16_0095
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Influenza
Keywords: Influenza; health care workers; nosocomial; asymptomatic; France
MeSH Terms: conditions — Influenza, Human | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health-care workers (Experimental): Health-care workers recruited in the study will have blood sampling and naso-pharyngeal bottle-brush sampling
  Interventions: Biological: Blood sampling; Other: Nasal swab

INTERVENTIONS:
Biological: Blood sampling
Other: Nasal swab

SUMMARY:
Although clinical presentation of influenza is often symptomatic, asymptomatic cases also occur. The knowledge of the incidence of asymptomatic influenza among healthcare workers is very important because of the risk of cross-transmission to hospitalized patients. The principal objective of the study is to estimate the incidence of symptomatic and asymptomatic influenza among healthcare workers in short-stay wards. The results of this study will lead to a better understanding of the burden of asymptomatic influenza among healthcare workers and might be used as an argument to increase influenza vaccine coverage among healthcare workers.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer health-care workers
* Working in the following wards: short-stay, inpatient (including ICU) and emergency

Exclusion Criteria:

* Presence of influenza symptoms at enrolment
* Programmed absence (maternity leave, vacation, etc.)
* Administrative agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2016-10-04 (Actual); Primary Completion 2017-03-21 (Actual); Study Completion 2017-03-21 (Actual)

PRIMARY OUTCOMES:
Incidence of influenza cases | 6 months after inclusion
  Incidence of asymptomatic and symptomatic influenza per 1000 days at risk among healthcare workers

SECONDARY OUTCOMES:
Fraction of asymptomatic influenza cases | 6 months after inclusion
  Fraction of asymptomatic influenza cases among patients with confirmed influenza infection (seroconversion)
Stratified incidence ratios | 6 months after inclusion
  The objective is to compare the proportion of asymptomatic influenza among vaccinated and unvaccinated healthcare workers, stratified on the type of influenza virus , gender, age, and other covariates
Incidence of influenza-like illness | 6 months after inclusion
  The objective is to calculate the incidence of influenza-like illness without virological confirmation
proportion of health-care workers with Influenza vaccine coverage | 6 months after inclusion
  The objective is to estimate the vaccination coverage against influenza among health care workers
Number of sick-leave days per participating ward | 6 months after inclusion
  The objective is to estimate the professional impact of influenza in a population of healthcare workers

CONTACTS AND LOCATIONS:
Locations (1):
- Edouard Herriot Hospital; Department of Epidemiology, Hygiene and Public Health, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Benet T, Amour S, Valette M, Saadatian-Elahi M, Aho-Glele LS, Berthelot P, Denis MA, Grando J, Landelle C, Astruc K, Paris A, Pillet S, Lina B, Vanhems P; AFP Study Group. Incidence of Asymptomatic and Symptomatic Influenza Among Healthcare Workers: A Multicenter Prospective Cohort Study. Clin Infect Dis. 2021 May 4;72(9):e311-e318. doi: 10.1093/cid/ciaa1109. PMID 32750120